CLINICAL TRIAL: NCT05967598
Title: Effect of Transcutaneous Auricular Vagl Nerve Electrostimulation of Brainstem Structures in Early and Late Parkinson's Disease Patients - an fMRI Study
Brief Title: Effect of taVNS of Brainstem Activation in Early and Late Parkinson's Disease Patients - an fMRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Vovk, Principal investigator, University of Ljubljana
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 012052/2020-2
Record Dates: First submitted 2023-04-05; First posted 2023-08-01 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Neurologic Disorder
Keywords: Parkinson disease; taVNS; transcutaneous auricular vagal nerve stimulation; fMRI; brainstem ROI analysis
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: 40 participants with the diagnosis of PD patients aged > 45 years will be included. Patients will be recruited from the outpatient and inpatient clinics. PD will be diagnosed according to the UK PD Society Brain Bank criteria: the investigators aim to include 20 patients with early-stage and 20 patients with late-stage PD. Each participant will complete 1 visit at the MRI scanning facility, during which they will complete 3 blocks of 8min block design fMRI. During each block they will receive a different kind of stimulation (taVNS25, taVNS100, xVNS; see detailed description).
  The effect will be compared within each group (early and advanced patients) and between groups (early vs advanced PD patients).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Before the experiment the stimulation threshold (i.e. current) for each stimulation (taVNS25 and taVNS100) will be assessed by a third person.
  The participant will be told, that the investigators are comparing the effect of 3 different stimulation types and that each will be delivered at a different intensity.
  The order of stimulation will be randomised across the 3 fMRI slots by a third person and the stimulation type will be noted in a separate log file.
  The outcomes assessor will be blinded to the stimulation type until the end of the analysis process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- taVNS100 in advanced PD patients (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 100Hz to advanced PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 100Hz
- taVNS25 in advanced PD patients (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 25Hz to advanced PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 25Hz
- xVNS in advanced PD patients (Placebo Comparator): The electrode will be placed in the left cyma conchae however no electrical current will be applied to advanced PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Sham cyma conchae stimulation
- taVNS100 in early PD patients (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 100Hz to early PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 100Hz
- taVNS25 in early PD patients (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 25Hz to early PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 25Hz
- xVNS in early PD patients (Placebo Comparator): The electrode will be placed in the left cyma conchae however no electrical current will be applied to early PD patients. Participants will complete an 8 minute block design fMRI block.
  Interventions: Device: Sham cyma conchae stimulation

INTERVENTIONS:
Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 100Hz — Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold at 100Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment
  Other Names: taVNS100
  Arms: taVNS100 in advanced PD patients; taVNS100 in early PD patients
Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 25Hz — Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold at 25Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment.
  Other Names: taVNS25
  Arms: taVNS25 in advanced PD patients; taVNS25 in early PD patients
Device: Sham cyma conchae stimulation — The electrode will be placed at the cymba conchae location, however no electrical current will be applied. All other experimental conditions will be the same as for the active taVNS stimulation.
  Other Names: xVNS
  Arms: xVNS in advanced PD patients; xVNS in early PD patients

SUMMARY:
This is a randomised, within-subject, double-blinded, placebo-controlled study to assess the fMRI correlates of central nervous system (CNS) response to taVNS in early vs late-stage Parkinsons disease (PD), at two different frequencies. Forty PD patients will be included: twenty patients with early-stage (Hoehn and Yahr stage (HY) 1-2) and twenty patients with late-stage (HY 3-4) PD. Each patient will undergo one stimulation session, where they will receive active taVNS at 100 Hz (taVNS100), taVNS at 25Hz (taVNS25) or will have positioned electrodes without stimulation (xVNS). The order of taVNS100, taVNS25 and xVNS will be randomized between subjects. The session will include (1) xVNS and taVNS; (2) MRI and fMRI and (3) heart rate and breathing rate monitoring. Clinical assessment with the Movement Disorder Society-Unified Parkinson's Disease Rating Scale will be done before the session.

DETAILED DESCRIPTION:
Each participant will complete 1 visit, where the investigators will first assess the MDS-UPDRS score, afther that the sesnsitivity threasholds for taVNS at 25Hz and taVNS at 100Hz will be assessed. The Nemos® electrode for taVNS will be positioned in the left cymba conchae with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs. taVNS25 will be applied at 25Hz and taVNS100 will be applied at 100Hz. The sensory threshold will be assessed for each frequency and in the MRI scanner a pulse intensity of 0,1mA above the perceptual threshold will be applied.

After that the participant will be escorted to the MRI scanner where the MRI-safe electrode will be positioned in the left cymba conchae. The participant will be instructed to hold their head still during the complete experiment and that they will receive 3 different electrical stimulation types during 3 separate sessions. They will be further instructed that a black dot that will appear on the screen before each stimulation session and that they should fix their gaze on the dot. The instructions will be repeated before each BOLD MRI session.

MRI will be performed at the Center for Clinical physiology at the Medical faculty in Ljubljana (Center za klinično fiziologijo; CKF), using a 3T Philips Achieva 3TX dStream (Best, The Netherlands).

The investigators will acquire high-resolution T1-weighted and T2-weighted (0.7 x 0.7 x 0.7 mm^3) volumes of the brain. The area of brainstem and cerebellum will be scanned using a T1-weighted spectral pre-saturation with inversion recovery (SPIR) sequence to enhance the contrast of neuromelanin structures (and better delineate LC). The three structural scans will be interspaced with 3 time slots, containing three 8 minutes long block design blood oxygen level-dependent (BOLD MRI; fMRI) sessions (~1.75mm^3 isometric voxel). During each fMRI slot participants will receive a different type of stimulation (taVNS,25, taVNS100 and xVNS). While the participant will receive electrical stimulation during taVNS25 and taVNS100, there will be no current applied during xVNS. To reduce any carryover effect the investigators will randomise the order of the 3 fMRI sessions. The order of stimulation will not be revealed until the automated data and statistical analysis.

The timeline of the complete imaging session would be as follows: Survey scan - Slot 1 - T1 - Slot 2 - T2 - Slot 3 - neuromelanin sequence. The session should last up to 60 min. During this time the investigators will monitor heart rate and breathing rate remotely.

For the analysis T1-weighted images will be first segmented into grey, white and cerebrospinal fluid (CSF) tissue compartments using DARTEL, implemented in SPM12. This also provides spatial normalization and co-registration to the standard MNI space. Images from other modalities will first be co-registered to T1-weighted structural scans and next to the MNI template as secondary images using the identical transform algorithm. From the fMRI data the investigators will analyse (i) brainstem activation patterns (ROI analysis); and (ii) block design connectivity between nucleus tractus solitarii and central nervous system (CNS) structures and locus coeruleus and CNS stuctures. fMRI analyses will be done with Analysis of Functional NeuroImages (AFNI) tools.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease according to the UK PD Society Brain Bank criteria
* ability to walk independently for at least 2 minutes
* cognitive impairment that might prevent cooperation during tests
* stable antiparkinsonian medications during the previous 1 month

Exclusion Criteria:

* medication resistant rest tremor or dyskinesias
* history of seizures
* implanted medical devices or metal implants
* pregnancy
* claustrophobia
* fixed or severe kyphosis
* any conditions that would prevent our patients from lying still for 1 hour in a supine position (i.e. muscle pain, degenerative joint diseases…).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Comparison of Brainstem activation pattern on fMRI (ROI analysis) during taVNS compared to xVNS | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Block-design fMRI analysis will be performed on brainstem ROIs to assess activation in neuromodulatory brainstem nuclei during taVNS compared with xVNS using the tools of the AFNI program. Final analysis will be performed on group level.
Comparison of Functional connectivity pattern on fMRI (block design) of nucleus tractus solitarii and the rest of the nervous system during taVNS compared to xVNS | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Functional connectivity (fMRI, block design) between the nucleus tractus solitarii (NTS) and the rest of the central nervous system will be analysed with AFNI Context-Dependent Correlation Analysis to determine whether taVNS produces a different pattern of connectivity compared with xVNS.
Comparison of Functional connectivity pattern on fMRI (block design) of locus coeruleus (LC) and the rest of the nervous system during taVNS compared to xVNS | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Functional connectivity pattern (fMRI, block design) between the nucleus locus coeruleus (LC) and the rest of the central nervous system will be analysed with AFNI Context-Dependent Correlation Analysis to determine whether taVNS produces a different pattern of connectivity compared with xVNS.

SECONDARY OUTCOMES:
Comparison of Brainstem activation pattern on fMRI (ROI analysis) during taVNS25 compared to taVNS100 | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Block-design fMRI analysis will be performed on brainstem ROIs to assess activation in neuromodulatory brainstem nuclei during taVNS100 compared with taVNS25 using the tools of the AFNI program. Final analysis will be performed on group level.
Comparison of Functional connectivity pattern on fMRI (block design) of nucleus tractus solitarii and the rest of the nervous system during taVNS25 compared to taVNS100 | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Functional connectivity (fMRI, block design) between the nucleus tractus solitarii (NTS) and the rest of the central nervous system will be analysed with AFNI Context-Dependent Correlation Analysis to determine whether taVNS produces a different pattern of connectivity compared with xVNS.
Comparison of Functional connectivity pattern on fMRI (block design) of locus coeruleus (LC) and the rest of the nervous system during taVNS100 compared to taVNS25 | Only the online/acute effect measured during stimulation (time frame duration of 8 minutes per stimulation type) will be analysed.
  Functional connectivity pattern (fMRI, block design) between the nucleus locus coeruleus (LC) and the rest of the central nervous system will be analysed with AFNI Context-Dependent Correlation Analysis to determine whether taVNS100 produces a different pattern of connectivity compared with taVNS25.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Vovk, PhD, Principal Investigator — Medical Faculty, University of Ljubljana
Locations (1):
- Neurology Department, UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the anonymised data with researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon request after study publication
Access Criteria: Data will be shared with researchers upon reasonable request